CLINICAL TRIAL: NCT06461338
Title: Acupuncture for Enhancing the Effect of Immunotherapy in Advanced NSCLC: a Pilot Study
Brief Title: Acupuncture for Enhancing Immunotherapy in Advanced NSCLC：a Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023YFC3503303
Record Dates: First submitted 2024-06-10; First posted 2024-06-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer; Non-Small-Cell Lung Carcinoma
Keywords: Non-Small Cell Lung Cancer; Acupuncture; Immune Checkpoint Inhibitors; Effect; Safety
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture for 4 times every 3 weeks (one cycle of ICIs combined with chemotherapy) for 12 weeks (4 cycles of ICIs combined with chemotherapy)
  Interventions: Procedure: acupuncture
- Sham acupuncture (Sham Comparator): Sham acupuncture for 4 times every 3 weeks (one cycle of ICIs combined with chemotherapy) for 12 weeks (4 cycles of ICIs combined with chemotherapy)
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: acupuncture — Acupuncture at Neiguan(PC6), Zhongwan (CV12), Guanyuan (CV 4), Baihui (DU20), Yintang (GV29), combined with electro-acupuncture at Zusanli(ST36), and Sanyinjiao (SP-6).
  Arms: Acupuncture
Procedure: Sham acupuncture — Sham acupuncture at Neiguan(PC6), Zhongwan (CV12), Guanyuan (CV 4), Baihui (DU20), Yintang (GV29), combined with sham electro-acupuncture at Zusanli(ST36), and Sanyinjiao (SP-6).
  Arms: Sham acupuncture

SUMMARY:
This multicentre, randomized controlled trial evaluates the effect and safety of integrating acupuncture with immunotherapeutic sensitization in treating NSCLC. Participants will be randomly assigned to undergo either acupuncture or sham acupuncture concurrent with the initial four cycles of standard ICIs combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Has a histologically-confirmed or cytologically confirmed diagnosis of stage IIIB or IV NSCLC.
2. PD-L1 TPS<50%
3. EGFR/ALK wild-type
4. Has not received prior systemic treatment for advanced NSCLC. For patients who received preoperative neoadjuvant chemotherapy or postoperative adjuvant chemotherapy or radical chemoradiotherapy, if the disease progresses occurred one six months after the last treatment, they can be enrolled. Patients who received targeted therapy or immunotherapy can not be enrolled.
5. Has a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
6. Age≥18 years
7. Has a life expectancy of at least 3 months
8. Has measurable disease
9. Has adequate organ function
10. Voluntarily enrolled into the study, sign the informed consent form and have good compliance

Exclusion Criteria:

1. Unable to complete baseline assessments
2. Expected to receive radiotherapy within the next 4 cycles
3. With a combination of serious primary diseases of the heart, cerebrovascular, hepatic, renal, and hematopoietic systems
4. With dementia, neurological disorders, mental retardation, or language impairment, and pregnant or breastfeeding women
5. Combined autoimmune diseases, hematologic disorders, or long-term use of hormones or immunosuppressive drugs
6. Combined with a primary tumor from other sites
7. Had participated in any other clinical trial within the prior 3 months
8. Has known history of Human Immunodeficiency Virus (HIV) or solid organ transplantation
9. With legal incapacity
10. With skin breakdown at the acupuncture point that interferes with treatment
11. With a pacemaker
12. With a fear of acupuncture
13. Had received acupuncture treatment within 6 weeks
14. Has known active Hepatitis B
15. Has interstitial lung disease or a history of pneumonitis that required oral of IV glucocorticoids to assist with management
16. Has fever (>38°C) or clinically significant infection within 1 week prior to enrolment
17. Has active tuberculosis or indications of severe or uncontrolled systemic diseases
18. With a bleeding tendency, and receiving thrombolytics or anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Progress free survival defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 5 years.
  Overall survival is defined as the time until death due to any cause
Objective response rate | Through study completion, an average of 3 years.
  Objective response rate is defined as the proportion of patients achieving complete (iCR/CR) or partial (iPR/PR) response according to iRECIST or RECIST V.1.1 criteria
Disease control rate | Through study completion, an average of 3 years.
  Disease control rate is determined by the percentage of patients who achieve CR, PR, or SD as defined by iRECIST or RECIST V.1.1 criteria. This encompasses all instances of CR, PR, and SD (CR + PR + SD).
Duration of response | Through study completion, an average of 3 years.
  Duration of response is assessed only in patients achieving CR, PR, or nPR and was defined as the time from first assessment showing CR, PR, or nPR to earliest date of either PD or death.
Quality of life evaluation | At the baseline, day 8 of Cycle 1-4 (each cycle is 21 days), and day 1 of Cycle 5 (each cycle is 21 days), up to approximately 6 months.
  According to the requirements of European Organisation for Research and Treatment of Cancer-quality of life core questionnaire (EORTC QLQ-C30)/Lung cancer 13 items (LC13), the scoring results of each field of the scale were recorded in CRF. The score of this questionnaire ranges between 1 and 4. The higher score indicates the worse quality of life.
Symptom evaluation | At the baseline, day 8 of Cycle 1-4 (each cycle is 21 days), and day 1 of Cycle 5 (each cycle is 21 days), up to approximately 6 months.
  According to the requirements of Lung cancer symptom scale (LCSS), the scoring results of each field of the scale were recorded in CRF. The score of this questionnaire ranges between 0 and 10. The higher score indicates the worse symptom.

OTHER OUTCOMES:
Next-generation sequencing | At the baseline and the date of first documented progression, up to approximately 36 months.
  Biopsy/surgery samples were examined histopathologically and for reptarenavirus RNA by qRT-PCR and metagenomic NGS.
  Genetic testing of tissue samples was performed by NGS.
Cytometry by time-of-flight | At the baseline and the date of first documented progression, up to approximately 36 months.
  Cells were analyzed using a CyTOF mass cytometer
Tumor markers | At the baseline and the date of first documented progression, up to approximately 36 months.
  Detection of tumor markers including serum carcinoembryonic antigen (CEA), neuron-specific enolase (NSE), squamous cell carcinoma (SCC), carbohydrate antigen 125 (CA125) and cytokeratin 19 fragment (CyFRA21-1).
Pro-inflammatory index | At the baseline and the date of first documented progression, up to approximately 36 months.
  Pro-inflammatory index were measured from the peripheral blood.
The traditional Chinese medicine syndrome evaluation | At the baseline, the end of Cycle 2 (each cycle is 21 days), and day 1 of Cycle 5 (each cycle is 21 days), up to approximately 6 months.
  The data related to Chinese medicine syndrome types will be extracted, including symptoms and signs, tongue, pulse, and other syndrome information.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, M.D., Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (3):
- China (3):
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine., Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Jiangsu Provincial Hospital of Chinese Medicine, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided